CLINICAL TRIAL: NCT01720160
Title: Barostim HOPE4HF Study
Brief Title: BAROSTIM® Hope for Heart Failure Study
Acronym: HOPE4HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 360032-001
Record Dates: First submitted 2012-10-29; First posted 2012-11-02 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure
Keywords: Systolic Heart Failure; Congestive Heart Failure; Reduced left ventricular ejection fraction; HFrEF
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Device (Experimental): 1) BAROSTIM NEO System and 2) standard of care medical management therapy for heart failure (American Heart Association [AHA] / American College of Cardiology [ACC] guidelines), including drugs (determined by the patient's physician). Drug types include: Loop Diuretics, Thiazide Diuretics, Potassium-sparing Diuretics, Sequential Nephron Blockade, ACE Inhibitors, ARBs, ARNI, Aldosterone Antagonists, Beta Blockers and Hydralazine and Isosorbide Dinitrate.
  Interventions: Device: BAROSTIM NEO® System; Other: Standard of care medical managment therapy for heart failure
- Medical Management (Active Comparator): Standard of care medical management therapy for heart failure (American Heart Association [AHA] / American College of Cardiology [ACC] guidelines), including drugs (determined by the patient's physician). Drug types include: Loop Diuretics, Thiazide Diuretics, Potassium-sparing Diuretics, Sequential Nephron Blockade, ACE Inhibitors, ARBs, ARNI, Aldosterone Antagonists, Beta Blockers and Hydralazine and Isosorbide Dinitrate.
  Interventions: Other: Standard of care medical managment therapy for heart failure

INTERVENTIONS:
Device: BAROSTIM NEO® System — Implant procedure
  Other Names: Neo® System
  Arms: Device
Other: Standard of care medical managment therapy for heart failure — Standard of care medical management therapy for heart failure (AHA/ACC guidelines), including drugs (determined by the patient's physician). Drug types include: Loop Diuretics, Thiazide Diuretics, Potassium-sparing Diuretics, Sequential Nephron Blockade, ACE Inhibitors, ARBs, ARNI, Aldosterone Antagonists, Beta Blockers and Hydralazine and Isosorbide Dinitrate.

SUMMARY:
The purpose of this clinical investigation is to assess the long-term safety and efficacy of the BAROSTIM NEO System in subjects currently participating in the BAROSTIM® HOPE4HF Trial (NCT01720160).

DETAILED DESCRIPTION:
A prospective, randomized study describing the safety and efficacy of the BAROSTIM NEO System in heart failure subjects with left ventricular ejection fraction equal to or less than 35 percent. Seventy two subjects were randomized; 32 to the medical management arm and 40 to the device arm (38 implanted, 2 withdrawn). The study closed to new enrollments on January 31, 2014. Subjects are in long-term follow-up and are required to have at least one annual visit. During the visit, there will be a physical assessment, a review of medications and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Actively participating in the BAROSTIM HOPE4HF Study and currently implanted with the BAROSTIM NEO device with the device turned ON.
* Have signed a revised approved informed consent form for continued participation in this study.

Exclusion Criteria:

• Treating physician decision that the subject should not continue with therapy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2012-11; Primary Completion 2015-05 (Actual); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Heart failure metric improvements from baseline | 12 months
  To describe changes in measures compared to baseline.
System and procedure related adverse events | 6 months
  To demonstrate the safety of the Neo system in a heart failure population.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zile, MD, Study Chair — Medical University of South Carolina; William Abraham, MD, Principal Investigator — Ohio State University; Fred Weaver, MD, Principal Investigator — University of Southern California; Faiez Zannad, MD, Principal Investigator — Inserm Centre d'Investigation, CHU de Nancy; JoAnn Lindenfield, MD, Principal Investigator — Vanderbilt Heart and Vascular Institute
Locations (23):
- United States (23):
  - Southwest Cardiovascular Associates, Mesa, Arizona
  - Arizona Heart Rhythm Research Center, Phoenix, Arizona
  - University of Southern California, Los Angeles, California
  - George Washington University, Washington D.C., District of Columbia
  - ACRC - Cardiology, Atlantis, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Advocate Medical Group, Naperville, Illinois
  - Cardiovascular Institute of the South, Houma, Louisiana
  - St Elizabeth's Medical Center, Brighton, Massachusetts
  - Mid-Michigan Medical Center Midland, Midland, Michigan
  - Cardiac & Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Ohio State University, Columbus, Ohio
  - Oklahoma Cardiovascular Research Group, Oklahoma City, Oklahoma
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Lonestar Heart Center, Amarillo, Texas
  - Wheaton Franciscan Healthcare, Milwaukee, Wisconsin
  - Aspirus Heart & Vascular Institute, Wausau, Wisconsin

REFERENCES:
- [Result] Abraham WT, Zile MR, Weaver FA, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Little WC. Baroreflex Activation Therapy for the Treatment of Heart Failure With a Reduced Ejection Fraction. JACC Heart Fail. 2015 Jun;3(6):487-496. doi: 10.1016/j.jchf.2015.02.006. Epub 2015 May 14. PMID 25982108
- [Derived] Halbach M, Abraham WT, Butter C, Ducharme A, Klug D, Little WC, Reuter H, Schafer JE, Senni M, Swarup V, Wachter R, Weaver FA, Wilks SJ, Zile MR, Muller-Ehmsen J. Baroreflex activation therapy for the treatment of heart failure with reduced ejection fraction in patients with and without coronary artery disease. Int J Cardiol. 2018 Sep 1;266:187-192. doi: 10.1016/j.ijcard.2018.04.075. Epub 2018 Apr 21. PMID 29705650
- [Derived] Zile MR, Abraham WT, Weaver FA, Butter C, Ducharme A, Halbach M, Klug D, Lovett EG, Muller-Ehmsen J, Schafer JE, Senni M, Swarup V, Wachter R, Little WC. Baroreflex activation therapy for the treatment of heart failure with a reduced ejection fraction: safety and efficacy in patients with and without cardiac resynchronization therapy. Eur J Heart Fail. 2015 Oct;17(10):1066-74. doi: 10.1002/ejhf.299. Epub 2015 Jun 10. PMID 26011593